CLINICAL TRIAL: NCT01954446
Title: A Novel Non-interfering Arterial Blood Pressure Monitoring Device
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The investigational devices need alterations before validation
Sponsor: Sense A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: DK011
Record Dates: First submitted 2013-05-29; First posted 2013-10-01 (Estimated); Last update posted 2013-10-01 (Estimated); Status verified 2013-09

CONDITIONS: Hypertension; Hypotension; Healthy
MeSH Terms: conditions — Hypertension; Hypotension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ContiPress vs. 3M (Experimental): ContiPress vs. 3M passive and during exercise
  Interventions: Device: 3M; Device: ContiPressTM
- ContiPress vs. Mobil-O-Graph (Experimental): ContiPress vs. Mobil-O-Graph passive, then oscillometric passive, then oscillometric for 24 hrs every 15 mins.
  Interventions: Device: 3M; Device: ContiPressTM; Device: Mobil-O-Graph

INTERVENTIONS:
Device: 3M — Conventional measuring of BP
Device: ContiPressTM — New way of measuring BP - ContiPressTM
  Investigational device
Device: Mobil-O-Graph — 2 different devices for oscillometric measurement of BP
  Arms: ContiPress vs. Mobil-O-Graph

SUMMARY:
The primary purpose of this investigation is to validate the performance and safety of the Investigational Device (ID) against a validated and legally cleared device for measuring Blood Pressure (BP). The secondary purpose is to validate the performance of the ID over a period of 24 hours against a validated and legally cleared device for Ambulatory Blood Pressure Monitoring (ABPM).

DETAILED DESCRIPTION:
The clinical investigation is conducted as a controlled (subject as own control), prospective, randomised, comparative investigation in a population with a representative spread of BPs to ensure that the ID performs as good as current marketed and approved devices. The study will be conducted in compliance with the International Standard ANSI/AAMI/ISO 81060-2 - Non-invasive sphygmomanometers - Clinical validation of automated measurement type.

This clinical investigation will enrol up to 96 male and female subjects to ensure the recording of 85/35 evaluable datasets in accordance with the ANSI/AAMI/ISO standard [11]. All measurements will be paired and falls into 2 categories: Auscultatory measurements as gold standard reference, oscillometric measurements for clinical practise reference and further validation of ambulatory monitoring and pulse shape measurements.

ELIGIBILITY:
Inclusion Criteria:

* At least 30% of the subjects must be males (n=29)
* At least 30% of the subjects must be female (n=29)
* Age ≥ 18 years old
* Limb size circumference ≥ 17 cm
* Blood pressure distribution:
* At least 25 % of the subjects should be hypertensive
* At least 5 % of the subjects should be hypotensive

Exclusion Criteria:

* Breached skin
* Acknowledged pregnancy
* Pacemaker
* Diagnosed cardiac arrhythmia (tachycardia, bradycardia, atrial/ventricular fibrillation)
* Implanted metal in upper limb:

  * Elbow prosthesis
  * Shoulder prosthesis
  * Metal screws
  * Bone plates
  * Metal chips
  * Surgical clips
  * Implantable Cardiac Defibrillator (ICD)
  * Cardiac Resynchronization Therapy - Defibrillator (CRT-D)
  * Premature ventricular contractions (PVC)
  * Premature arterial contractions (PAC)
  * Sensitivity or allergy towards adhesives
* Presence of an arterial-venous shunt
* Recent axillary node dissection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-04; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Accuracy of measurement | Up to 4 months
  The reference measurements are compared with the measurements made by the investigational device

SECONDARY OUTCOMES:
Skin irritation | Up to 4 months
  After removal of each investigational device the skin is assessed. Also participants are instructed to report any skin irritation to investigator

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Olsen, Prof. MD, Principal Investigator — Odense University Hospital